

# **Tool Revision History:**

| Version Number | Version Date | Summary of Revisions Made |
|---|---|---|
| 1.0 | 20 DEC 2017 | Original version |
| 2.0 | 05 JAN 2017 | Amended version |
| 3.0 | 18 JAN 2018 | Reflects change in HBV screening to account for vaccination |
| 4.0 | 05 MAY 2018 | Removes exclusion for combined organ recipients |
| 5.0 | 05 JUL 2018 | Modifies wording of donor HBV exclusion criterion |
| 6.0 | 19 JUL 2018 | Increase enrollment target to 20 patients |
| 7.0 | 27 JUL 2018 | Specifies risks with regard to transmitting HCV infection |
| 8.0 | 28 AUG 2018 | Directly states participant inclusion ages as 18 and older |



# A SINGLE-CENTER PILOT STUDY OF THE USE OF HEPATITIS C POSITIVE DONORS FOR HEPATITIS C NEGATIVE HEART TRANSPLANT RECIPIENTS WITH POST-TRANSPLANT TREATMENT OF HEPATITIS C VIREMIA WITH MAVYRET

| Principal Investigator: | Alex Reyentovich, MD |
|---|---|
| | Associate Professor of Medicine |
| | Clinical Director, Heart Failure Program |
| | Medical Director, Heart Transplant and Ventricular Assist Device |
| | Program |
| | The Leon H. Charney Division of Cardiology, NYU Langone Health |
| | 530 First Avenue, Suite-9N |
| | New York, NY 10016 |
| | 646-501-0119 |
| | Alex.Reyentovich@nyumc.org |
| Additional Investigators: | Co-investigators: |
| | Nader Moazami, MD (Nader.Moazami@nyumc.org) |
| | Bonnie Lonze, MD PHD (Bonnie.Lonze@nyumc.org) |
| | Ira Jacobson, MD (Ira.Jacobsom@nyumc.org) |
| | Claudia Gidea, MD (Claudia.Gidea@nyumc.org) |
| NYULMC Study Number: | S17-01775 |
| Funding Sponsor: | None |
| IND/IDE Number: | None |
| Regulatory Sponsor: | None |
| Study Product: | Mavyret (glecaprevir/pibrentasvir) |
| Study Product Provider: | AbbVie, Inc., North Chicago, IL |
| ClinicalTrials.gov Number | Submitted; pending review for assignment of registration number |

Initial version: 20 December 2017
Amended: 05 January 2018
Amended: 18 January 2018
Amended: 05 May 2018
Amended: 05 July 2018
Amended: 19 July 2018
Amended: 27 July 2018
Amended: 28 August 2018

Version:8.0

# **Statement of Compliance**

This study will be conducted in accordance with the Code of Federal Regulations on the Protection of Human Subjects (45 CFR Part 46), 21 CFR Parts 50, 56, 312, and 812 as applicable, any other applicable US government research regulations, and institutional research policies and procedures. The International Conference on Harmonisation ("ICH") Guideline for Good Clinical Practice ("GCP") (sometimes referred to as "ICH-GCP" or "E6") will be applied only to the extent that it is compatible with FDA and DHHS regulations. The Principal Investigator will assure that no deviation from, or changes to the protocol will take place without prior agreement from the sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants. All personnel involved in the conduct of this study have completed Human Subjects Protection Training.

Study number: s17-01775


# **Table of Contents**

| S | TATEMENT OF COMPLIANCE | III |
|---|---|---|
| L | IST OF ABBREVIATIONS | VIII |
| Ρ | ROTOCOL SUMMARY | 1 |
| S | CHEMATIC OF STUDY DESIGN | 2 |
| 1 | KEY ROLES | 3 |
| 2 | INTRODUCTION, BACKGROUND INFORMATION AND SCIENTIFIC RATIO | |
| | <ul> <li>2.1 BACKGROUND INFORMATION AND RELEVANT LITERATURE</li> <li>2.2 NAME AND DESCRIPTION OF THE INVESTIGATIONAL AGENT</li> </ul> | |
| | 2.2.1 Preclinical Data | |
| | 2.2.2 Clinical Data to Date | |
| | 2.2.3 Dose Rationale (if applicable) | |
| | 2.3 RATIONALE | |
| | 2.4 POTENTIAL RISKS & BENEFITS | |
| | 2.4.2 Known Potential Benefits | |
| 3 | | |
| | 3.1 PRIMARY OBJECTIVE | |
| | 3.2 SECONDARY OBJECTIVES | |
| 4 | STUDY DESIGN AND ENDPOINTS | |
| _ | 4.1 DESCRIPTION OF STUDY DESIGN | |
| | 4.2 STUDY ENDPOINTS | |
| | 4.2.1 Primary Study Endpoints | |
| | 4.2.2 Secondary Study Endpoints | 7 |
| 5 | STUDY ENROLLMENT AND WITHDRAWAL | 7 |
| | 5.1 INCLUSION CRITERIA | 7 |
| | 5.2 EXCLUSION CRITERIA | |
| | 5.3 VULNERABLE SUBJECTS | |
| | 5.4 STRATEGIES FOR RECRUITMENT AND RETENTION | |
| | 5.5 Duration of Study Participation | |
| | 5.6 TOTAL NUMBER OF PARTICIPANTS AND SITES | 9 |
| | 5.7 PARTICIPANT WITHDRAWAL OR TERMINATION | |
| | 5.7.1 Reasons for Withdrawal or Termination | |
| | 5.7.2 Handling of Participant Withdrawals or Termination | |
| 6 | STUDY AGENT | |
| J | | |
| | 6.1 STUDY AGENT(S) AND CONTROL DESCRIPTION | |

| | udy number: s | 17-01775 | Page v |
|---|---|---|---|
| Ve | ersion:8.0<br>6.1.2 | Formulation, Appearance, Packaging, and Labeling | 10 |
| | 6.1.3 | Product Storage and Stability | |
| | 6.1. <del>4</del> | Preparation | |
| | 6.1. <del>5</del> | Dosing and Administration | |
| | 6.1.6 | Route of Administration | |
| | 6.1.7 | Dose Adjustments/Modifications/Delays | |
| | 6.1.8 | Duration of Therapy | |
| | 6.1.9 | Tracking of Dose | |
| | | JDY AGENT ACCOUNTABILITY PROCEDURES | |
| 7 | | PROCEDURES AND SCHEDULE | |
| • | | | |
| | | JDY PROCEDURES/EVALUATIONS | |
| | 7.1.1 | Study Specific Procedures | 11 |
| | 7.1.2 | Standard of Care Study Procedures | |
| | | ORATORY PROCEDURES/EVALUATIONS | |
| | 7.2.1 | Clinical Laboratory Evaluations | |
| | 7.2.2 | Other Assays or Procedures | |
| | 7.2.3 | Specimen Preparation, Handling, and Storage | |
| | 7.2.4 | Specimen Shipment | 13 |
| | 7.3 STU | JDY SCHEDULE | 13 |
| | 7.3.1 | Screening | |
| | 7.3.2 | Enrollment/Baseline | |
| | 7.3.3 | Intermediate Visits | 14 |
| | 7.3.4 | Final Study Visit - for all patients | 16 |
| | 7.3.5 | Withdrawal/Early Termination Visit | 17 |
| | 7.3.6 | Unscheduled Visit | 17 |
| | 7.4 Co | NCOMITANT MEDICATIONS, TREATMENTS, AND PROCEDURES | 17 |
| | 7.4.1 | Precautionary Medications, Treatments, and Procedures | 17 |
| | 7.5 PR | OHIBITED MEDICATIONS, TREATMENTS, AND PROCEDURES | 17 |
| | 7.6 RES | SCUE MEDICATIONS, TREATMENTS, AND PROCEDURES | 18 |
| | | RTICIPANT ACCESS TO STUDY AGENT AT STUDY CLOSURE | |
| 8 | ASSES | SMENT OF SAFETY | 18 |
| | 8.1 SPE | ECIFICATION OF SAFETY PARAMETERS | 10 |
| | 8.1.1 | Definition of Adverse Events (AE) | |
| | 8.1.1 | | |
| | 8.1.2<br>8.1.3 | Definition of Serious Adverse Events (SAE) | |
| | | Definition of Unanticipated Problems (UP) | |
| | 8.2 CLA<br>8.2.1 | ASSIFICATION OF AN ADVERSE EVENT | |
| | _ | Severity of Event | |
| | 8.2.2 | Relationship to Study Agent | |
| | 8.2.3 | Expectedness | |
| | | E PERIOD AND FREQUENCY FOR EVENT ASSESSMENT AND FOLLOW-UP | |
| | | PORTING PROCEDURES – NOTIFYING THE IRB | |
| | 8.4.1 | Adverse Event Reporting | 21 |
| | 8.4.2 | Serious Adverse Event Reporting | |
| | 8.4.3 | Unanticipated Problem Reporting | |
| | 8.4.4 | Reporting of Pregnancy | |
| | 8.5 STU | JDY HALTING RULES | 22 |

| Study nu<br>Version:8 | mber: s17-01775 Page | iv ; |
|---|---|---|
| 8.6 | SAFETY OVERSIGHT | . 22 |
| 9 CI | INICAL MONITORING | . 22 |
| 10 | STATISTICAL CONSIDERATIONS | . 23 |
| 10.1 | STATISTICAL AND ANALYTICAL PLANS (SAP) | . 23 |
| 10.2 | STATISTICAL HYPOTHESES | . 23 |
| 10.3 | | |
| 10.4 | | |
| | 9.4.1 General Approach<br>9.4.2 Analysis of the Primary Efficacy Endpoint(s) | |
| _ | 1.4.2 Analysis of the Secondary Endpoint(s) | |
| _ | 1.4.4 Safety Analyses | |
| 10 | 1.4.5 Adherence and Retention Analyses | |
| | 2.4.6 Baseline Descriptive Statistics | |
| | 1.4.7 Planned Interim Analysis | |
| | 9.4.8 Multiple Comparison/Multiplicity9.4.9 Tabulation of Individual Response Data | |
| _ | SAMPLE SIZE | |
| | SOURCE DOCUMENTS AND ACCESS TO SOURCE DATA/DOCUMENTS. | |
| | QUALITY ASSURANCE AND QUALITY CONTROL | |
| 13 | ETHICS/PROTECTION OF HUMAN SUBJECTS | . 26 |
| 13.1 | ETHICAL STANDARD | |
| 13.2 | | |
| 13.3 | Informed Consent Process | . 26 |
| | 2.3.1 Consent/Assent and Other Informational Documents Provided | |
| | articipants | |
| 13.4 | | |
| | DATA HANDLING AND RECORD KEEPING | |
| 14.1 | Data Collection and Management Responsibilities | 27 |
| 14.2 | | |
| 14.3 | | |
| 14.4 | PUBLICATION AND DATA SHARING POLICY | . 28 |
| 15 | STUDY FINANCES | . 29 |
| 15.1 | FUNDING SOURCE | . 29 |
| 15.2 | Costs to the Participant | |
| 16 | STUDY ADMINISTRATION | . 29 |

ATTACHMENTS ...... 32

**17** 

18

19

| Study no | umber: s17-01775 | Page vii |
|----------|--------------------|----------|
| Version: | 8.0 | |
| 20 | SCHEDULE OF EVENTS | 35 |


#### **List of Abbreviations**

AE Adverse Event/Adverse Experience

CFR Code of Federal Regulations

CRF Case Report Form

DHHS Department of Health and Human Services

DSMB Data and Safety Monitoring Board

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

HBV Hepatitis B Virus
HCV Hepatitis C Virus

HIV Human Immunodeficiency Virus

ICF Informed Consent Form

ICH International Conference on Harmonisation

IRB Institutional Review Board
MOP Manual of Procedures

N Number (typically refers to participants)

NIH National Institutes of Health

OHRP Office for Human Research Protections
OHSR Office of Human Subjects Research

PHS Public Health Service
PI Principal Investigator
PMW Post-Mavyret weeks
POW Post-operative weeks
QA Quality Assurance
QC Quality Control

SAE Serious Adverse Event/Serious Adverse Experience

SOP Standard Operating Procedure
SVR Sustained virologic response

UNOS United Network for Organ Sharing

US United States

# **Protocol Summary**

| Protocol Summary | |
|---|---|
| Title | A single-center pilot study of the use of hepatitis C positive donors for hepatitis C negative heart transplant recipients with post-transplant treatment of hepatitis C viremia with Mavyret |
| Short Title | HCV positive heart donors |
| Brief Summary | Patients who are hepatitis C negative and are on the waiting list for a heart transplant will be enrolled. Study subjects will receive a heart transplant from a deceased donor who has tested positive for hepatitis C. Recipients will undergo surveillance for the development of hepatitis C viremia post-transplant. Those who develop viremia will be treated with an FDA-approved drug, Mavyret, which is a pan-genotypic hepatitis C treatment with a cure rate of over 98%. Treated patients will be monitored in order to ensure that cure of hepatitis C viremia with sustained virologic response has been achieved. |
| Phase | Pilot study |
| Objectives | To determine safety and efficacy of the strategy of transplantation of hearts from HCV positive donors (with or without evidence of active HCV viremia). To characterize the incidence of HCV viremia in recipients whose heart donors were HCV positive. For recipients who develop viremia, to characterize the time course of the development of viremia, and subsequent clearance of viremia after treatment with Mavyret. |
| Methodology | Open label, single treatment arm |
| Endpoint | Percentage of patients with sustained virologic response after treatment for HCV after heart transplant. Incidence of viremia after receiving a heart transplant from a donor who tests positive for hepatitis C. |
| Study Duration | Two years |
| Participant Duration | One year |
| Duration of IP administration | Eight weeks |
| Population | Adult patients active on the UNOS waiting list for a heart transplant |
| Study Sites | Single center (NYU Langone Hospital) |
| Number of participants | Ten patients |
| Description of Study<br>Agent/Procedure | The heart transplantation will be performed per standard of care techniques, and all post-transplant management of the transplanted organ, including immunosuppression, will be carried out per standard of care. The study-specific interventions will be surveillance for the development of hepatitis C viremia post-transplant, the treatment of viremia with an FDA-approved drug, and then surveillance for sustained virologic response post-treatment. |
| Reference Therapy | Not applicable |
| Key Procedures | Monitoring for transmission of hepatitis C after heart transplant, treatment of viremia if it develops, and monitoring for response to treatment. |
| Statistical Analysis | In this small pilot study, descriptive statistics will be used. |
| · | · |


# **Schematic of Study Design**




# 1 Key Roles

# **Principal Investigator**

Alex Reyentovich, MD
Associate Professor of Medicine
Clinical Director, Heart Failure Program
Medical Director, Heart Transplant and Ventricular Assist Device Program
The Leon H. Charney Division of Cardiology, NYU Langone Health
530 First Avenue, Suite-9N
New York, NY 10016



Nader Moazami, MD Professor of Surgery Surgical Director, Heart Transplantation and Mechanical Circulatory Support NYU Langone Cardiothoracic Surgery Associates 530 1st Avenue, Suite 9V New York, NY 10016

Bonnie Lonze, MD PhD Assistant Professor of Surgery Vice Chair for Research, NYU Langone Transplant Institute 403 E 34<sup>th</sup> St, 3<sup>rd</sup> Floor, New York, NY 10016

Ira Jacobson, MD Professor of Medicine Director, Hepatology NYU Langone Hepatology Associates 530 1<sup>st</sup> Avenue, Suite 4J New York, NY 10016

Claudia Gidea, MD Associate Director of VAD and Heart Transplant NYU Langone Cardiothoracic Surgery Associates 530 1<sup>st</sup> Avenue, Suite SK 9N New York, NY 10016


#### **Study Coordinators:**

Jennifer Pavone AGAGNP-BC Heart Failure/VAD/Transplant Program Manager NYU Langone Cardiothoracic Surgery Associates



#### **Research Coordinators:**

Elaina Weldon, MSN, ACNP-BC Transplant Research Nurse Practitioner NYU Langone Transplant Institute



Cecilia Deterville, MS, CCRC Senior Clinical Research Coordinator NYU Langone Transplant Institute



Gabriella Boulton, BA Associate Transplant Coordinator NYU Langone Transplant Institute



## 2.1 Background Information and Relevant Literature

In New York state, 2840 patients have received heart transplants since the year 2000. In that time, however 835 patients either died on the waiting list or became too sick for transplant [1]. Thus, for every 4 patients waitlisted in New York, one patient will die or become too sick for transplant before an organ becomes available. The shortage of organs available for heart transplantation directly results in loss of life.

At the same time, since 2000, in New York alone, 3,081 donor hearts were discarded because of donor history of HCV infection or exposure [2]. With the availability of new and well-tolerated direct-acting antiviral agents, cure rates for chronic HCV infection approach 100% [3]. Treatment of HCV naïve transplant recipients who develop donor-derived HCV infection post-transplant would be expected to be equally successful. Thus, if post-transplant antiviral treatment could enable HCV positive heart donors to be utilized for negative recipients, then the current donor pool has the potential to eliminate waitlist mortality.


There is, in fact, precedent for this as a viable strategy to narrow the gap between organ supply and demand. A recently study in which HCV positive donor kidneys were transplanted into HCV negative recipients demonstrated both excellent outcomes in terms of allograft function, and 100% HCV cure rates among the recipients [4]. Other ongoing and unpublished series of kidney transplant recipients [5] and of heart transplant recipients [6] have observed that only about 70% of HCV negative recipients who receive an organ from a HCV positive donor actually develop HCV viremia post-transplant. This is not surprising since the designation for HCV donor positivity by UNOS is a positive test for *either* anti-HCV antibody *or* HCV RNA. Donors who test positive for HCV antibody alone may have a falsely positive test, or may have had a prior exposure to HCV with subsequent virus clearance; in either scenario, there would be no risk of transmission of HCV infection to a recipient. It is estimated that 33% of donors designated as HCV positive are, in fact, non-viremic [7].

In this pilot study we propose utilizing HCV positive donors for HCV negative patients on the waiting list for a heart transplant at NYU Langone. We will propose careful early post-transplant surveillance for the development of HCV viremia. We anticipate that approximately one-third of the patients will not develop viremia, despite the donor designation HCV positive. We anticipate that two-thirds of patients will develop early post-transplant HCV viremia. These patients will be immediately treated with an FDA-approved anti-HCV therapy which we expect will cure the HCV.

Willingness to participate in this trial will afford patients quicker access to heart transplantation, and will have the potential to reduce waitlist mortality.

# 2.2 Name and Description of the Investigational Agent

Mavyret (glecaprevir/pibrentasvir)

Manufacturer: AbbVie, Inc., North Chicago IL

Mavyret is an FDA-approved, marketed drug clinically indicated for the treatment of HCV infection in patients without cirrhosis.

Its formulation is as an oral tablet containing two antiviral agents: glecaprevir and pibrentasvir. Glecaprevir is an inhibitor of the HCV NS3/4A protease which is essential for viral replication. Pibrentasvir is an inhibitor of the HCV NS5 protease which is necessary for RNA replication and virion assembly. Mavyret is active against all known strains of HCV.

#### 2.2.1 Preclinical Data

In vitro studies demonstrating efficacy of glecaprevir and pibrentasvir at preventing replication of all strains of HCV were published prior to the initiation of clinical trials for these agents. In vitro the two agents act synergistically and have high potency with low rates of resistance. [8]

#### 2.2.2 Clinical Data to Date

In Phase 3 clinical trials, 8 weeks of Mavyret therapy achieved high rates (98%) of SVR across all genotypyes (1-6) of HCV in patients with HCV infection without cirrhosis. Clinical trials involved over 2300 patients in 27 countries. Based on the results of clinical trials, the FDA approved Mayvret for use in the treatment of HCV (all strains) in patients without cirrhosis. (ClinicalTrials.gov identifiers:

NCT02651194, NCT02642432, NCT02640482, NCT02636595, NCT02604017, NCT02446717,

NCT02640157, NCT02243293) [9-14].

Included in the clinical trial populations were patients with severe renal impairment (stage 4 or 5 CKD). In this population Mavyret was found to be effective in achieving a high rate of SVR and no dosing adjustment was required [15].


#### 2.2.3 Dose Rationale (if applicable)

The dose used will be the standard dosing regimen for its FDA approved indication, three tablets taken once daily with food (total daily dose: glecaprevir 300mg and pibrentasvir 120mg)

#### 2.3 Rationale

There is a vast shortage of available organs for lifesaving heart transplants. Donors with history of HCV represent an unutilized source of organs that could potentially eliminate the current waiting list mortality. With the emergence of new, FDA approved treatments, HCV disease is now curable in nearly 100% of patients who contract it. By transplanting patients with HCV positive donor hearts, this study will offer the benefit of avoiding waiting list mortality, followed by treatment (with the expectation of cure) of HCV in the event of transmission.

#### 2.4 Potential Risks & Benefits

#### 2.4.1 Known Potential Risks

Risks of treatment failure: HCV mutation can lead to drug resistance and treatment failure. In patients administered Mavyret, the risk of this was 2% or less. For patients with treatment resistant HCV, rescue therapy with alternative agents can result in cure of up to 100% depending upon the genotype. Guidelines for the treatment of resistant HCV strains are published and updated regularly [16].

Risks of treatment intolerance: Over multiple clinical trials. the overall rate of medication related adverse events leading to permanent discontinuation prior to completion of an 8-week course of Mavyret therapy was 0.1% [17].

Risk of acute hepatitis C infection: Acute hepatitis C is asymptomatic in 66-75% of patients. The risks of acute HCV leading to fulminant hepatic failure are believed to be very low, however case reports of this do exist [18]. During the time that patients are acutely infected with hepatitis C infection, it is possible that patients could transmit infection to other individuals, if others individuals are exposed to the patient's blood. Family members who, for instance, assist patients with medical care such as diabetic blood sugar monitoring, could potentially be exposed to hepatitis C if they were to sustain a needlestick injury from a needle used by the patient. The risk of an infected individual transmitting hepatitis C via a needlestick exposure is approximately 5%. Patients in the study will be counseled to use caution to prevent blood exposure to other individuals and will be asked to notify the study team immediately if they believe any individuals were exposed to their blood during the duration of the study participation.

Risk of chronic hepatitis C infection: Patients who prove refractory to all therapy including rescue therapy and develop persistent viremia are at risk to develop chronic HCV infection which has the potential to cause cirrhosis/end-stage liver disease, the potential for the need for liver transplantation and/or death. We expect our treatment failure rate in this study to be 0%, therefore we expect the risk of chronic HCV infection to be 0%. In the event of a treatment failure, the risks of developing chronic HCV must be considered. It is estimated that approximately 15-30% of patients with chronic HCV develop cirrhosis/end-stage liver disease over 20-30 years [19]. This risk should be compared to the risk of death on the heart transplant waiting list. The reported one-year mortality for a waitlisted patient without a transplant is as high 26.7% [20].

The efficacy of HCV treatment with Mavyret is high (98%). The efficacy of rescue therapies approaches 100%. Even in the event of a treatment failure, the risk of cirrhosis and liver disease secondary to chronic HCV are low. We believe that the survival benefit of receiving an earlier heart transplant, by accepting an organ from a HCV positive donor, far outweighs the risks of HCV exposure and possible treatment failure.


## 2.4.2 Known Potential Benefits

The benefit of this study is the ability to obtain a lifesaving heart transplant rather than risk death while waiting on the list for a HCV negative organ.

# 3 Objectives and Purpose

#### 3.1 Primary Objective

This pilot feasibility study is being conducted to determine safety and efficacy of the strategy of transplantation of hearts from HCV positive donors (with or without evidence of active HCV viremia) into HCV negative recipients on the NYU Langone Health heart transplant waiting list, with subsequent anti-HCV therapy to treat infection in the recipient.

# 3.2 Secondary Objectives

Secondary objectives will include characterization of the incidence of HCV viremia in recipients whose heart donors were HCV positive.

For those who develop viremia we will also characterize the time course of the development of viremia, and subsequent clearance of viremia after treatment.

# 4 Study Design and Endpoints

# 4.1 Description of Study Design

This will be an open-label, single arm, single center trial of the use of HCV positive heart donors for HCV negative recipients, followed by treatment of HCV infection in recipients who develop viremia.

#### 4.2 Study Endpoints

#### 4.2.1 Primary Study Endpoints

The primary endpoint will be percentage of patients with sustained virologic response after treatment for HCV after heart transplant.

This endpoint was chosen as primary because it will enable us to evaluate the safety of transient exposure to HCV at the time of heart transplantation. The expectation is that all patients who develop HCV viremia will achieve SVR (cure) following treatment with Mavyret.

#### 4.2.2 Secondary Study Endpoints

Secondary endpoints will include:

1-year patient survival rates in HCV negative heart recipients who receive a heart transplant from a HCV positive donor.

Incidence of acute HCV viremia among HCV negative recipients who receive a heart transplant from a HCV positive donor.

These endpoints will enable us to assess the risks associated with this approach to heart transplantation and will allow us to better understand the risks of this approach to risks associated with remaining on the waiting list for a HCV-negative organ offer.

# 5 Study Enrollment and Withdrawal

#### 5.1 Inclusion Criteria

In order to be eligible to participate in this study, an individual must meet all of the following criteria:


1. Listed for heart transplant at NYU Langone Health (including candidates listed for dual organs)

- 2. Able to travel to the NYU Langone Health for routine post-transplant visits and study visits for a minimum of 6 months after transplantation
- 3. No active illicit substance abuse
- 4. Weight at least 50kg
- 5. Women of childbearing potential must agree to use birth control in accordance with Mycophenolate Risk Evaluation and Mitigation Strategy (REMS) after transplant due to the increased risk of birth defects and/or miscarriage
- 6. Both men and women must agree to use at least one barrier method after transplant to prevent any secretion exchange
- 7. Able and willing to provide informed consent
- 8. Age 18 years old and older

Furthermore, the deceased donors from whom the organs will be procured must meet the following criteria:

- 1. Detectable HCV RNA by nucleic acid test (NAT) or positive anti-HCV antibody
- 2. Donor heart meets standard NYU Langone Health clinical criteria for procurement

#### 5.2 Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

- 1. HIV positive
- 2. HCV RNA positive or history of previously treated HCV
- 3. Evidence of active Hepatitis B infection or on active antiviral treatment for HBV
- 4. Pregnant or nursing (lactating) women
- 5. Use of strong CYP3A inducers

Furthermore, the deceased donors from whom the organs will be procured will be excluded if they meet any of the following criteria:

- 1. Confirmed HIV positive
- 2. Evidence of active HBV infection
- 3. Known previously failed treatment for HCV

#### 5.3 Vulnerable Subjects

Vulnerable subjects will not be eligible for enrollment.

#### 5.4 Strategies for Recruitment and Retention

Recruitment of patients will occur during routine evaluation visits to determine candidacy for a heart transplant at NYU Langone Heath. Patients will be informed of the option to enroll in this study, and if interested, detailed information pertaining to the risks and benefits of the trial will be provided.

The signing of the acknowledgment to consider participation in the study will occur in the outpatient clinic. No additional information about potential candidates will be collected to determine interest or candidacy for this trial than would otherwise be normally collected as per standard of care for evaluation for a heart transplant.

Written informed consent for actual enrollment in the study will occur in the inpatient setting once a viable organ offer has been identified and the patient is admitted for potential transplantation.

The target sample size will be 20 patients.


## 5.4.1 Use of DataCore/Epic Information for Recruitment Purposes

This study may utilize EPIC to identify subjects.

Any recruitment information sent by email will utilize Send Safe email.

Potential subjects will already be known to the study team as they will be under their care as candidates and/or waitlist registrants for heart transplant. The study team will conduct an in person consultation with the patients to explain the study as well as discuss the risks, benefits, and alternatives

Approved recruitment language will be used to communicate the reason they are being contacted and subjects will be asked if they are interested in participating in this specific study. Should the potential subjects agree, the study team will provide the subjects with information regarding the next steps for participation.

If a subject requests information regarding opting out of further recruitment for all research, subjects will be directed to contact research-contact-optout@nyumc.org or 1-855-777-7858.

#### 5.5 Duration of Study Participation

Duration of participation is expected to be 12 months.

#### 5.6 Total Number of Participants and Sites

20 patients are expected to be enrolled and transplanted. No sites outside of NYULMC will enroll patients.

# 5.7 Participant Withdrawal or Termination

#### 5.7.1 Reasons for Withdrawal or Termination

Participants are free to withdraw from participation in the study at any time upon request. An investigator may terminate participation in the study if:

- Any clinical adverse event (AE), laboratory abnormality, or other medical condition or situation
  occurs such that continued participation in the study would not be in the best interest of the
  participant
- The participant meets an exclusion criterion (either newly developed or not previously recognized) that precludes further study participation

#### 5.7.2 Handling of Participant Withdrawals or Termination

Discontinuation of the study agent is not anticipated as this will place patients at risk to develop acute or chronic HCV. For patients who do elect to discontinue the study agent Mavyret due to intolerance or SAEs/AEs, the following steps will be taken:

Hepatology consultation to guide management, which could include:

Continued surveillance for evidence of HCV viremia in patients who had cleared their viremia Conversion to an alternate HCV treatment that is able to be tolerated by the patient

#### 5.8 Premature Termination or Suspension of Study

This study may be temporarily suspended or prematurely terminated if there is sufficient reasonable cause. Written notification, documenting the reason for study suspension or termination, will be provided by the suspending or terminating party to the Principal Investigator. If the study is prematurely terminated or suspended, the PI will promptly inform the IRB and will provide the reason(s) for the termination or suspension.

Circumstances that may warrant termination or suspension include, but are not limited to:

- Determination of unexpected, significant, or unacceptable risk to participants
- Demonstration of efficacy that would warrant stopping


This material is the property of the NYU School of Medicine and Langone Medical Center. Do not disclose or use except as authorized in writing by the study sponsor


- Insufficient compliance to protocol requirements
- Data that are not sufficiently complete and/or evaluable
- Determination of futility

Study may resume once concerns about safety, protocol compliance, data quality is addressed and satisfy the IRB and DSMB.

#### 6 Study Agent

# 6.1 Study Agent(s) and Control Description

Mavyret is available in tablet form. The single tablet contains two active agents: glecaprevir (100nmg) and pibrentasvir (40mg).

No IND is required here as this is an FDA-approved agent for the treatment of HCV infection. The drug is marketed and will be available through the pharmacy. In accordance with FDA Guidelines, we attest that this study meets all of the following exemption criteria and that no IND is required:

- Mavyret is lawfully marketed in the United States
- This investigation is not intended to be reported to the FDA in support of a new indication for Mavyret
- This investigation is not intended to support a change in marketing for Mavyret
- This investigation does not involve a route of administration, dosing change, or patient population change compared to what is FDA-approved for Mavyret
- This investigation will be conducted in compliance with the NYULMC IRB review and consenting requirements
- This investigation is not intended to promote or commercialize the product Mavyret.

Detailed documentation of the above FDA Guidelines is also uploaded as an attachment in Research Navigator.

# 6.1.1 Acquisition

These agents are FDA approved and will be obtained from the NYULMC pharmacy via standard procedure for medication ordering.

## 6.1.2 Formulation, Appearance, Packaging, and Labeling

This is an open label study and the drug will appear as it provided directly from the manufacturer. The tablets are pink, oblong-shaped, film-coated, and debossed with "NXT" on one side. The drug will be packed in the standard manufacturer's packing and all standard and package inserts will be retained.

# 6.1.3 Product Storage and Stability

Mavyret is dispensed from the manufacturer in a 4-week (monthly) or an 8-week carton. Each weekly carton contains seven daily dose wallets. Each monthly carton contains four weekly cartons. Each 8-week carton contains 2 monthly cartons. Each child resistant daily dose wallet contains three 100 mg/40 mg glecaprevir/pibrentasvir tablets. Storage is at room temperature.

#### 6.1.4 Preparation

The drug is a tablet for oral ingestion. No preparation is required.

# 6.1.5 Dosing and Administration

The dose will be three tablets taken at one time, once daily with a meal. The standard duration of therapy is daily administration for 8-weeks.


#### 6.1.6 Route of Administration

Oral

# 6.1.7 Dose Adjustments/Modifications/Delays

No dose adjustments are anticipated. Subjects will be counseled as to the importance of strict adherence to the medication regimen. Subjects will be advised to notify the study team of any missed or delayed doses. If a dose is missed and less than 18 hours have elapsed since the scheduled time, patients will be instructed to take the missed dose with the next meal and resume the regular schedule the following day. If a dose is missed and more than 18 hours have elapsed since the scheduled time, then the patients will be instructed not to take the missed dose, but to resume the regular schedule the next day.

#### 6.1.8 Duration of Therapy

The duration of therapy will be 8-weeks.

#### 6.1.9 Tracking of Dose

While in the hospital, any doses will be given by nursing staff and accountability will be maintained in the electronic medical record. Once outpatient, patients will attend regularly scheduled clinic appointments for routine care following a heart transplant and medication review will occur on each of these visits to ensure that the medication is being taken properly. Laboratory testing for HCV will be performed as described. Clearance of HCV and SVR will serve as clinical evidence that the mediation is being taken properly.

# 6.2 Study Agent Accountability Procedures

For therapy that is initiated during the inpatient hospitalization post-transplant, the NYU Langone pharmacy will dispense the medication and it will be given to the patient by the bedside nurse. For outpatient therapy the drug will be distributed to the study subjects together with the standard of care medications they will require after a heart transplant. The drug is supplied in either 4-week or 8-week batches. Completion of the course will leave no remaining doses. All the supplied product will be used.

#### 7 Study Procedures and Schedule

#### 7.1 Study Procedures/Evaluations

#### 7.1.1 Study Specific Procedures

Note that the medical history and medication history that pertains to candidacy for heart transplantation are considered standard of care procedures and evaluations for heart transplantation, and are not considered here. Patients are not considered candidates for this trial if there is any contraindication to their standard candidacy for a heart transplant. As such, procedures and evaluations specific to participation in this study include:

- Medical history to assess for any history of acute or chronic liver disease, and any prior infection with HCV, HBV, or HIV
- Medication history to assess for any potential interacting drugs including (amiodarone, statins, anti-epileptics, hormonal contraceptives, antipsychotics, recreational drugs, immunosuppressant drugs)
- Physical examination (height, weight, baseline blood pressure, heart rate, oxygen saturation, assess for absence of jaundice/scleral icterus, abdominal examination to assess for absence of hepatosplenomegaly, ascites, abdominal wall varices)
- Laboratory evaluations. Serum evaluation for HCV and HBV NAT testing. Serum evaluation for HCV HBV and HIV serologies, described in detail below.


 A discussion of if the results of any positive blood tests for HCV infection, and discussions of response to treatment once treatment has begun.

#### 7.1.2 Standard of Care Study Procedures

Heart transplantation and all associated procedures will be considered standard of care including: the transplant procedure itself and requisite intra-operative procedures and hemodynamic monitoring, post-operative ICU-level care, inpatient hospital unit care, outpatient post-operative care including, standard induction and maintenance immunosuppression, and standard post-transplant anti-infectious prophylaxis (anti-fungal, anti-pneumocystis, and anti-CMV prophylaxis).

## 7.2 Laboratory Procedures/Evaluations

## 7.2.1 Clinical Laboratory Evaluations

The following tests will be reviewed and recorded for patients who are included in the study but will be performed as standard of care for heart transplant recipients:

- Hematology: hemoglobin, hematocrit, white blood cells (WBC) with differential count, platelet count
- Biochemistry: sodium, potassium, CO2, BUN, creatinine, total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase
- Coagulation: INR
- **Pregnancy test**, usually to be done within 24 hours prior to study intervention and results must be available prior to administration of study product.
- HBV NAT testing: PCR test for detection and quantification of HBV viral load, an indicator of
  active HBV infection. These tests are performed as standard of care for patients who receive
  transplanted organs from a donor who is designated "PHS increased infectious risk." By
  definition, all HCV positive organ donors meet criteria for designation as PHS increased infectious
  risk.
- HBV serologic testing (HBsAb, HBsAg, HBcoreAb): serologic testing to evaluate for the
  presence of immunity to HBV or the evidence of prior infection with HBV. These tests are
  performed as standard of care for patients who receive transplanted organs from a donor who is
  designated "PHS increased infectious risk." By definition, all HCV positive organ donors meet
  criteria for designation as PHS increased infectious risk.
- HIV serologic testing (HIV1 and 2 antigen/antibody 4<sup>th</sup> gen): serologic testing to evaluate for the presence of HIV infection. These tests are performed as standard of care for patients who receive transplanted organs from a donor who is designated "PHS increased infectious risk." By definition, all HCV positive organ donors meet criteria for designation as PHS increased infectious risk.

The following tests will be performed specifically for purposes of this study:

HCV genotyping:

#### Hepatitis C Viral RNA, Genotype, LiPA®

Recipient testing for HCV genotyping will be ordered by standard ordering procedures through Epic as with all other tests.

- HCV NAT testing: PCR test for detection and quantification of HCV viral load
- HCV serologic testing: serologic evaluation for the presence of anti-HCV antibodies

# 7.2.2 Other Assays or Procedures




#### 7.2.3 Specimen Preparation, Handling, and Storage



See attached documents (Section 19) for detailed standard operating procedures for specimen processing, collection and shipping instructions from Quest Laboratories, as well as for the accreditation documentation for the Transplant Research Lab, where these specimens will be processed and stored.

#### 7.2.4 Specimen Shipment

Serum samples sent to Quest Laboratories will be shipped frozen, according to collection and shipment instructions from Quest (see attachment in Section 19).

# 7.3 Study Schedule

#### 7.3.1 Screening

# Screening Visit (Day -365 to -1)

- Review medical history and perform physical examination to determine eligibility based on inclusion/exclusion criteria.
- Review medications history to determine eligibility based on inclusion/exclusion criteria.
- Collect blood to ensure that potential subjects have no evidence of current or prior infection with HCV, HBV, or HIV: HCV NAT and serologies, HBV NAT and serologies, HIV.
- Collect blood for documentation of pre-transplant liver function: hematology, biochemistry, coagulation
- Provide participants with detailed information about the study, in particular, conduct a detailed
  conversation of the risks and benefits of the trial. Risks discussed will include but not be limited
  to: risks of contracting treatment-resistant HCV and potential consequences of chronic HCV
  infection. Benefits discussed will include but not be limited to: shortened time to heart
  transplantation, and minimizing of the chance of death on the waiting list while waiting for a HCV
  negative organ offer. A Fact Sheet outlining the basic objectives, procedures, risks and benefits
  will be provided to patients.
- Obtain written acknowledgement of willingness to participate in study and receipt of Fact Sheet.

#### 7.3.2 Enrollment/Baseline

#### Enrollment/Baseline Visit (Day -1 to 0)


• Organ offer for a HCV-positive donor heart is received. The donor inclusion criteria are reviewed to ensure all donor criteria are met.

- The organ offer and the opportunity to participate in the trial are discussed with the patient and if the patient accepts, the patient is then admitted to the hospital in preparation for heart transplant.
- Inclusion/exclusion criteria for the recipient are reviewed again
- Written informed consent to participate in the trial is obtained.
- Obtain urine pregnancy test from any woman participant of childbearing age.
- Record vital signs, results of examinations, other assessments.
- Collect blood for baseline hematology, biochemistry coagulation, HCV NAT and serologies, HBV NAT and serologies, and HIV serology.
- Heart transplant operation is performed as per standard of care techniques.
- Donor blood is acquired with the donor organ, and donor serum sent to Quest Laboratories for HCV genotyping (to be performed in parallel with the transplant). Donor serum is banked for repeat testing in the event of indeterminate genotyping results.

#### 7.3.3 Intermediate Visits

For the schedules below, the following time-post-event designations will be used:

**POW** (Post-operative week) – refers to weeks following the transplant operation **PMW** (Post-Mavyret treatment week) – refers to weeks following the initiation of Mavyret therapy

All patients post-transplant will enter the Surveillance Phase which will entail weekly screening for the development of HCV viremia post-transplant for 8 weeks. Time in the surveillance phase is measured in reference to the transplant itself, in POW. Patients who never develop HCV viremia during the Surveillance Phase will transition to the No Transmission schedule detailed below. Time in the No Transmission arm is measured in reference to the transplant itself, in POW.

Patients who develop detectable HCV viremia during the Surveillance Phase will immediately exit the Surveillance Phase and enter the Mavyret Treatment arm schedule as detailed below. Time in the Mayvret Treatment arm is measured in reference to the date that Mavyret treatment was initiated, in PMW.

# SURVEILLANCE PHASE SCHEDULE OF EVENTS

#### POW1 (+/- 1 day)

- In person visit, record vital signs
- · Record standard of care labs: hematology, biochemistry, coagulation
- Collect study labs: HCV NAT

#### POW2 (+/- 2 days)

- In person visit, record vital signs
- Record standard of care labs: hematology, biochemistry, coagulation
- Collect study labs: HCV NAT

#### POW3 (+/- 3 days)

- Record standard of care labs: hematology, biochemistry, coagulation
- Collect study labs: HCV NAT

#### POW4 (+/- 5 days)

- In person visit, record vital signs
- Record standard of care labs: hematology, biochemistry, coagulation, HBV serologies and NAT, HIV serologies
- Collect study labs: HCV NAT


## POW5 (+/- 5 days)

• Record standard of care labs: hematology, biochemistry, coagulation

Collect study labs: HCV NAT

## POW6 (+/- 5 days)

• Record standard of care labs: hematology, biochemistry, coagulation

Collect study labs: HCV NAT

#### POW7 (+/- 5 days)

Record standard of care labs: hematology, biochemistry, coagulation

Collect study labs: HCV NAT

# POW8 (+/- 5 days)

Record vital signs

Record standard of care labs: hematology, biochemistry, coagulation,

Collect study labs: HCV NAT and serology

# NO TRANSMISSION ARM SCHEDULE OF EVENTS

#### POW12 (+/- 7 days)

In person visit, record vital signs

 Record standard of care labs: hematology, biochemistry, coagulation, HBV serologies and NAT, HIV serologies

Collect study labs: HCV NAT and serology

## POW16 (+/- 7 days)

Record standard of care labs: hematology, biochemistry, coagulation

Collect study labs: HCV NAT and serology

# POW20 (+/- 7 days)

Record standard of care labs: hematology, biochemistry, coagulation

Collect study labs: HCV NAT and serology

#### POW24 (+/- 14 days): INTERIM ASSESSMENT AT 6-months post-transplant

In person visit, record vital signs

Record standard of care labs: hematology, biochemistry, coagulation

Collect study labs: HCV NAT and serology

#### MAVYRET TREATMENT ARM SCHEDULE OF EVENTS

## PMW0 (+/- 5 days of determination of HCV viremia)

Initiate Mavyret therapy (daily dosing x 8 weeks)

• In person visit, record vital signs

#### PMW1 (+/- 1 day)

Record standard of care labs: hematology, biochemistry, coagulation

Collect study labs: HCV NAT and serology

#### PMW2 (+/- 2 day)

Record standard of care labs: hematology, biochemistry, coagulation

Collect study labs: HCV NAT and serology

#### PMW3 (+/- 3 day)

Record standard of care labs: hematology, biochemistry, coagulation


This material is the property of the NYU School of Medicine and Langone Medical Center. Do not disclose or use except as authorized in writing by the study sponsor


· Collect study labs: HCV NAT and serology

#### PMW4 (+/- 5 day)

- In person visit, record vital signs
- Record standard of care labs: hematology, biochemistry, coagulation, HBV serologies and NAT, HIV serologies
- Collect study labs: HCV NAT and serology

#### PMW5 (+/- 5 day)

- Record standard of care labs: hematology, biochemistry, coagulation
- Collect study labs: HCV NAT and serology

## PMW6 (+/- 5 day)

- Record standard of care labs: hematology, biochemistry, coagulation
- Collect study labs: HCV NAT and serology

# PMW7 (+/- 5 day)

- Record standard of care labs: hematology, biochemistry, coagulation
- Collect study labs: HCV NAT and serology

#### PMW8 (+/- 5 day)

- In person visit, record vital signs
- Confirm completion of Mavyret treatment course
- Record standard of care labs: hematology, biochemistry, coagulation
- Collect study labs: HCV NAT and serology

# PMW9 (+/- 5 day)

- Record standard of care labs: hematology, biochemistry, coagulation
- Collect study labs: HCV NAT and serology

#### PMW10 (+/- 5 day)

- Record standard of care labs: hematology, biochemistry, coagulation
- Collect study labs: HCV NAT and serology

#### PMW11 (+/- 5 day)

- Record standard of care labs: hematology, biochemistry, coagulation
- Collect study labs: HCV NAT and serology

## PMW12 (+/- 5 day)

- Record standard of care labs: hematology, biochemistry, coagulation
- Collect study labs: HCV NAT and serology

#### PMW16 (+/- 5 day)

- Record standard of care labs: hematology, biochemistry, coagulation
- Collect study labs: HCV NAT and serology

# POW24 (+/- 14 days): INTERIM ASSESSMENT AT 6-months post-transplant

- In person visit, record vital signs
- Record standard of care labs: hematology, biochemistry, coagulation
- Collect study labs: HCV NAT and serology

# 7.3.4 Final Study Visit - for all patients


## POW52 (+/- 14 days): FINAL ASSESSMENT AT 12-months post-transplant

• In person visit, record vital signs

 Record standard of care labs: hematology, biochemistry, coagulation, HBV serologies and NAT, HIV serologies

Collect study labs: HCV NAT and serology

# 7.3.5 Withdrawal/Early Termination Visit

Early withdrawal will be strongly discouraged for patients and the need to complete the entire follow-up course will be discussed with patients prior to enrolling in the study. Concern for the ability to follow-up will constitute exclusion from entry into the study.

For patients who do not develop HCV viremia post-transplant early withdrawal from the study will mean incomplete surveillance for the possible development of HCV. The importance of this screening will be discussed in detail with any person who elects to discontinue the follow-up.

Patients who develop HCV viremia and begin treatment, who elect to terminate treatment prior to the completion of the course will be counseled that this constitutes a risk for the development of chronic HCV and potential liver disease and/or liver failure in the future. Patients who elect to terminate therapy will be referred to a hepatologist for long-term follow-up and surveillance after HCV infection/exposure.

In general, we do not anticipate that there will be any withdrawal or early termination from the patients who enroll in this study. Because these patients will have had a heart transplant and maintaining a heart transplant generally requires close follow-up both for monitoring of graft function and for monitoring of immunosuppression, in general this is a very low risk group of patients to be lost to follow-up.

#### 7.3.6 Unscheduled Visit

Patients who undergo heart transplantation are expected to have a need for unscheduled visits depending on their clinical course. Unscheduled visits that pertain directly to the trial (i.e. due to reactions or intolerances to Mavyret, due to illness associated with acute HCV infection, HCV resistances) will occur as clinically appropriate and any AEs/SAEs will be documented as described below.

# 7.4 Concomitant Medications, Treatments, and Procedures

The subjects will receive concomitant medications which would otherwise be given as standard of care for patients undergoing a heart transplant.

All concomitant prescription medications taken during study participation will be recorded on the case report forms (CRFs). For this protocol, a prescription medication is defined as a medication that can be prescribed only by a properly authorized/licensed clinician. Medications to be reported in the CRF are concomitant prescription medications, over-the-counter medications and non-prescription medications.

#### 7.4.1 Precautionary Medications, Treatments, and Procedures

Treatment with amiodarone, digoxin, atorvastatin, lovastatin, simvastatin, pravastatin, rosuvastatin, flucastatin, pitavastatin requires special consideration and possible dosing adjustments in patients receiving Mavyret and the use of these medications will be discussed by the study team and any dose adjustment plan documented in the CRF.

# 7.5 Prohibited Medications, Treatments, and Procedures

Treatment with atazanavir, darunavir, lopinavir, ritonavir, efavirenz, rifampin, cyclosporine, ethinyl estradiol-containing oral contraceptives, carbamazepine, dabigatran, St. John's wort will not be permitted.


## 7.6 Rescue Medications, Treatments, and Procedures

In the event that a subject fails to achieve SVR with Mavyret, rescue therapy with other marketed agents approved for the treatment of HCV will be administered. The rescue treatment will be determined based on genotyping and resistance testing, and the choice of drug(s) used will be prescribed under the direction of a transplant hepatologist and/or transplant infectious diseases physician.

#### 7.7 Participant Access to Study Agent at Study Closure

Not applicable

#### 8 Assessment of Safety

#### 8.1 Specification of Safety Parameters

## 8.1.1 Definition of Adverse Events (AE)

An **adverse event** (AE) is any symptom, sign, illness or experience that develops or worsens in severity during the course of the study. Intercurrent illnesses or injuries should be regarded as adverse events. Abnormal results of diagnostic procedures are considered to be adverse events if the abnormality:

- results in study withdrawal
- is associated with a serious adverse event
- · is associated with clinical signs or symptoms
- · leads to additional treatment or to further diagnostic tests
- is considered by the investigator to be of clinical significance

## 8.1.2 Definition of Serious Adverse Events (SAE)

#### **Serious Adverse Event**

Adverse events are classified as serious or non-serious. A serious adverse event is any AE that is:

- fatal
- life-threatening
- · requires or prolongs hospital stay
- · results in persistent or significant disability or incapacity
- a congenital anomaly or birth defect
- an important medical event

Important medical events are those that may not be immediately life threatening, but are clearly of major clinical significance. They may jeopardize the subject, and may require intervention to prevent one of the other serious outcomes noted above. For example, drug overdose or abuse, a seizure that did not result in in-patient hospitalization, or intensive treatment of bronchospasm in an emergency department would typically be considered serious.

All adverse events that do not meet any of the criteria for serious should be regarded as **non-serious adverse events**.

#### 8.1.3 Definition of Unanticipated Problems (UP)

#### **Unanticipated Problems Involving Risk to Subjects or Others**

Any incident, experience, or outcome that meets all of the following criteria:

• <u>Unexpected in nature, severity, or frequency</u> (i.e. not described in study-related documents such as the IRB-approved protocol or consent form, the investigators brochure, etc.)


This material is the property of the NYU School of Medicine and Langone Medical Center. Do not disclose or use except as authorized in writing by the study sponsor


• Related or possibly related to participation in the research (i.e. possibly related means there is a reasonable possibility that the incident experience, or outcome may have been caused by the procedures involved in the research)

• <u>Suggests that the research places subjects or others at greater risk of harm</u> (including physical, psychological, economic, or social harm).

#### 8.2 Classification of an Adverse Event

## 8.2.1 Severity of Event

For AEs not included in the protocol defined grading system, the following guidelines will be used to describe severity.

- Mild Events require minimal or no treatment and do not interfere with the participant's daily
  activities
- **Moderate** Events result in a low level of inconvenience or concern with the therapeutic measures. Moderate events may cause some interference with functioning.
- **Severe** Events interrupt a participant's usual daily activity and may require systemic drug therapy or other treatment. Severe events are usually potentially life-threatening or incapacitating.

# 8.2.2 Relationship to Study Agent

The clinician's assessment of an AE's relationship to study is part of the documentation process, but it is not a factor in determining what is or is not reported in the study. If there is any doubt as to whether a clinical observation is an AE, the event should be reported. All AEs must have their relationship to study agent assessed. In a clinical trial, the study product must always be suspect. To help assess, the following guidelines are used.

- Related The AE is known to occur with the study agent, there is a reasonable possibility that the study agent caused the AE, or there is a temporal relationship between the study agent and event. Reasonable possibility means that there is evidence to suggest a causal relationship between the study agent and the AE.
- Not Related There is not a reasonable possibility that the administration of the study agent
  caused the event, there is no temporal relationship between the study agent and event onset, or
  an alternate etiology has been established.

For all collected AEs, the clinician who examines and evaluates the participant will determine the AE's causality based on temporal relationship and his/her clinical judgment. The degree of certainty about causality will be graded using the categories below.

- Definitely Related There is clear evidence to suggest a causal relationship, and other possible
  contributing factors can be ruled out. The clinical event, including an abnormal laboratory test
  result, occurs in a plausible time relationship to drug administration and cannot be explained by
  concurrent disease or other drugs or chemicals. The response to withdrawal of the drug
  (dechallenge) should be clinically plausible. The event must be pharmacologically or
  phenomenologically definitive, with use of a satisfactory rechallenge procedure if necessary.
- **Probably Related** There is evidence to suggest a causal relationship, and the influence of other factors is unlikely. The clinical event, including an abnormal laboratory test result, occurs within a reasonable time after administration of the drug, is unlikely to be attributed to concurrent disease or other drugs or chemicals, and follows a clinically reasonable response on withdrawal (dechallenge). Rechallenge information is not required to fulfill this definition.
- Possibly Related There is some evidence to suggest a causal relationship (e.g., the event occurred within a reasonable time after administration of the trial medication). However, other


factors may have contributed to the event (e.g., the participant's clinical condition, other concomitant events). Although an AE may rate only as "possibly related" soon after discovery, it can be flagged as requiring more information and later be upgraded to "probably related" or "definitely related," as appropriate.

- Unlikely to be related A clinical event, including an abnormal laboratory test result, whose temporal relationship to drug administration makes a causal relationship improbable (e.g., the event did not occur within a reasonable time after administration of the trial medication) and in which other drugs or chemicals or underlying disease provides plausible explanations (e.g., the participant's clinical condition, other concomitant treatments).
- Not Related The AE is completely independent of study drug administration, and/or evidence
  exists that the event is definitely related to another etiology. There must be an alternative,
  definitive etiology documented by the clinician.

# 8.2.3 Expectedness

The Principal Investigator will be responsible for determining whether an AE is expected or unexpected. An AE will be considered unexpected if the nature, severity, or frequency of the event is not consistent with the risk information previously described for the study agent.

# 8.3 Time Period and Frequency for Event Assessment and Follow-Up

The occurrence of an AE or SAE may come to the attention of study personnel during study visits and interviews of a study participant presenting for medical care, or upon review by the DSMB. All AEs including local and systemic reactions not meeting the criteria for SAEs will be captured on the appropriate CRF. Information to be collected includes event description, time of onset, clinician's assessment of severity, relationship to study product (assessed only by those with the training and authority to make a diagnosis), and time of resolution/stabilization of the event. All AEs occurring while on study must be documented appropriately regardless of relationship. All AEs will be followed to adequate resolution.

Any medical condition that is present at the time that the participant is screened will be considered as baseline and not reported as an AE. However, if the study participant's condition deteriorates at any time during the study, it will be recorded as an AE. UPs will be recorded in the data collection system throughout the study.

Changes in the severity of an AE will be documented to allow an assessment of the duration of the event at each level of severity to be performed. AEs characterized as intermittent require documentation of onset and duration of each episode.

The PI will record all reportable events with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation. At each study visit, the investigator will inquire about the occurrence of AE/SAEs since the last visit. Events will be followed for outcome information until resolution or stabilization.

All unresolved adverse events should be followed by the investigator until the events are resolved, the subject is lost to follow-up, or the adverse event is otherwise explained. At the last scheduled visit, the investigator should instruct each subject to report any subsequent event(s) that the subject, or the subject's personal physician, believes might reasonably be related to participation in this study. The investigator should notify the study sponsor of any death or adverse event occurring at any time after a subject has discontinued or terminated study participation that may reasonably be related to this study. The sponsor should also be notified if the investigator should become aware of the development of cancer or of a congenital anomaly in a subsequently conceived offspring of a subject that has participated in this study.


## 8.4 Reporting Procedures - Notifying the IRB

# 8.4.1 Adverse Event Reporting

All AEs will be recorded in AE CRFs by a member of the study team. AEs will be recorded within 3 business days of the study team being made aware of the AE. The relationship of the AE to the study interventions will be noted by the PI. AEs that are deemed definitely related or probably related to the study interventions will be reported to the IRB and the DSMB within 3 days of their designation as such. The DSMB will determined the need for an emergency meeting between the DSMB and the study team (see safety oversight below). AEs that are deemed unrelated or not likely related to the study interventions will be recorded on CRFs as described above and will be reviewed at quarterly DSMB safety review meetings, and at annual review by the IRB.

# 8.4.2 Serious Adverse Event Reporting

All SAEs will be recorded in SAE CRFs by a member of the study team. SAEs will be recorded within 3 business days of the study team being made aware of the SAE. The relationship of the SAE to the study interventions will be noted by the PI. SAEs that are both unexpected and deemed related to the study interventions will be reported to the IRB and the DSMB within 24 hours of the PI designation as such. The DSMB will determined the need for an emergency meeting between the DSMB and the study team (see safety oversight below) or whether these can be reviewed at quarterly meetings. SAEs that are deemed unrelated or not likely related to the study interventions will be recorded on CRFs, will be reported to IRB and DSMB within 3 days of their designation as such and will be reviewed at quarterly DSMB safety meetings.

# 8.4.3 Unanticipated Problem Reporting

Incidents or events that meet the OHRP criteria for UPs require the creation and completion of an UP report form. It is the site investigator's responsibility to report UPs to their IRB and notify the DSMB. The UP report will include the following information:

- Protocol identifying information: protocol title and number, PI's name, and the IRB project number;
- A detailed description of the event, incident, experience, or outcome;
- An explanation of the basis for determining that the event, incident, experience, or outcome represents an UP;
- A description of any changes to the protocol or other corrective actions that have been taken or are proposed in response to the UP.

To satisfy the requirement for prompt reporting, UPs will be reported using the following timeline:

- UPs that are SAEs will be reported to the IRB within 3 days the investigator becoming aware of the event.
- Any other UP will be reported to the IRB within 3 days of the investigator becoming aware of the problem.

# 8.4.4 Reporting of Pregnancy

If any pregnancy occurs in a study subject, the PI will be notified immediately and the IRB will be notified within 3 days of discovery of the pregnancy. No data regarding safety or efficacy of Mavyret in pregnant women are available. Standard of care medications utilized for heart transplant recipients have known contraindications in pregnancies therefore any pregnancies will need to be managed as per standard of care with the heart transplant team. Counseling of pregnant subjects with regard to the risks of continuing versus discontinuing Mavyret will occur with patients once counseling with regard to the contraindications of the standard of care transplant medications has occurred.


## 8.5 Study Halting Rules

Further enrollment of study subjects will be halted under the following conditions:

- Any patient death occurs and is deemed related to the intervention
- Any SAE deemed related to acute HCV infection occurs
- Any SAE deemed related to Mavyret occurs

The PI will inform the IRB and the DSMB within 24 hours of any of these events. The DSMB and study team will convene an emergency meeting as described below. The DSMB will provide recommendations for proceeding with any further enrollment. Patients who are already enrolled and receiving Mavyret treatment will continue to receive treatment unless the DSMB determines that an alternate course of therapy should be pursued for already-enrolled subjects.

#### 8.6 Safety Oversight

It is the responsibility of the Principal Investigator to oversee the safety of the study. This safety monitoring will include careful assessment and appropriate reporting of adverse events as noted above, as well as the construction and implementation of a site data and safety-monitoring plan. Medical monitoring will include a regular assessment of the number and type of serious adverse events.

Safety oversight will be under the direction of a DSMB. This DSMB committee for this study will be comprised of individuals with expertise in transplantation, hepatology, infectious diseases and the treatment of hepatitis C, and ethics. These individuals will be:

Arthur Caplan, PhD – Expert in medical ethics Nicole Ali, MD – Transplant nephrologist Stephen Pan, MD – Cardiologist Stuart Katz, MD – Cardiologist James Park, MD – Hepatologist Sapna Mehta, MD – Transplant infectious diseases

The DSMB Charter with specific outlines of DSMB roles and responsibilities is uploaded as a separate attachment in Research Navigator.

The DSMB will be notified of all AEs and SAEs as outlined above in 8.4.1 and 8.4.2. Regular meetings of the DSMB and the study team will occur on a quarterly basis to review non-emergent AEs and SAEs. The minimum group required to constitute an adequate DSMB-study team meeting will be (either in person or by teleconference): at least 4 of the DSMB members listed above, the PI, and at least one coinvestigator. At quarterly meetings the DSMB will evaluate cumulative participant safety data and make recommendations regarding the safe continuation of the study.

The DSMB and study team will meet on an emergency basis in the following instances:

- Any SAE occurs that is unexpected and deemed related to the study intervention
- Any unanticipated problem occurs that is both serious and deemed related to the study intervention
- Any treatment failure occurs or drug resistant HCV strain is identified, and a rescue plan with alternate therapy is required

Emergency meetings will occur within one business day of the above-described event occurring or being recognized. Any event that prompts an emergency DSMB-study team meeting will be reported to the IRB within 24 hours of the event occurring or being recognized.

## 9 Clinical Monitoring


Clinical site monitoring is conducted to ensure that the rights and well-being of human subjects are protected, that the reported trial data are accurate, complete, and verifiable, and that the conduct of the trial is in compliance with the currently approved protocol/amendment(s), with GCP, and with applicable regulatory requirement(s).

#### 10 Statistical Considerations

#### 10.1 Statistical and Analytical Plans (SAP)

As this is a single-arm observational study, no SAP will apply.

## 10.2 Statistical Hypotheses

We hypothesize that 100% of patients who develop HCV viremia will achieve SVR after completing an 8-week course of Mavyret treatment.

#### 10.3 Analysis Datasets

Subjects will be entered into a study subject dataset which includes de-identified information. This will include: donor and recipient demographic data, donor HCV NAT, serology, and genotyping information, and results of all recipient HCV NAT, serologic, and genotyping data obtained throughout the course of the study.

## 10.4 Description of Statistical Methods

Since the anticipated study population will be a small size, statistical analyses will be limited to descriptive statistics. For patients who develop post-transplant viremia we will be able to compare our HCV cure rates to those that are expected for patients who receive treatment with these agents for chronic HCV.

#### 10.4.1 General Approach

The study design will be single arm, open label. Descriptive statistics will include:

Incidence HCV viremia post-transplant (percentage)

Time course of exposure to development of clinically detectable viremia in those who develop viremia (median time to viremia with standard deviations)

Incidence of sustained clearance of HCV (cure) after treatment of viremia (percentage)

Time course of clearance of viremia after treatment initiation (median time to clearance with standard deviations)

Incidence of treatment failure/treatment resistant strains of HCV (percentage)

Characterization of distribution of HCV genotypes in patients who develop viremia (percentages)

Comparison of treatment failure rates to expected treatment failure rates for the treatments used (p value for significance will be set at p<0.05 and two-tailed t-test will be used)

#### 10.4.2 Analysis of the Primary Efficacy Endpoint(s)

The primary endpoint will be percentage of patients with sustained virologic response after treatment for HCV after heart transplant.

We expect that 100% of patients who are treated will achieve SVR. SVR will be defined as the absence of detectable HCV by NAT testing 3 months after the completion of the treatment course.

# 10.4.3 Analysis of the Secondary Endpoint(s)

Secondary endpoint #1: 1-year patient survival rates in HCV negative heart recipients who receive a heart transplant from a HCV positive donor.


This material is the property of the NYU School of Medicine and Langone Medical Center. Do not disclose or use except as authorized in writing by the study sponsor


Patients will have regular follow-up as standard of care for all heart transplant recipients. Patients survival will be readily apparent. Furthermore, all deaths of transplant recipients are required to be reported to UNOS.

Secondary endpoint #2: Incidence of HCV viremia among HCV negative recipients who receive a heart transplant from a HCV positive donor.

We will be measuring serial HCV NAT and serologic testing for a minimum of 6-months post-transplant. A patient will be considered to be viremic when a post-transplant HCV NAT test is positive. The incidence of viremia will be calculated as a percentage of the patients transplanted with a HCV-positive donor who develop HCV viremia by NAT testing.

#### 10.4.4 Safety Analyses

Safety concerns will be evaluated in real time. All AEs deemed to be related to the drug Mavyret will be evaluated by the PI. Any SAE deemed related to the drug Mavyret will be reported to the Monitoring committee within 3 days of PI notification of the event. Any AE or SAE deemed related to acute HCV infection will be reported to the Monitoring committee within 3 days of its determination. Any patient who is deemed a treatment failure (as defined by persistence of HCV viremia after completion of the full course of therapy) will be reported to the DSMB and the IRB within 3 days of its determination. A rescue course of therapy will be initiated under the direct guidance of a hepatologist and/or transplant infectious diseases specialist.

#### 10.4.5 Adherence and Retention Analyses

Adherence to the protocol will be assessed by the study team in direct conversations with the patients during routing visits, and will be assessed clinically by evaluation of HCV viral loads. Clearance of HCV will demonstrate adherence to the regimen. Failure to clear viremia will prompt more detailed direct patient inquiries regarding and will prompt an evaluation of possible treatment resistant strains of HCV as described elsewhere.

#### 10.4.6 Baseline Descriptive Statistics

In this study, no designed comparison groups will exist. The "No Transmission" arm and the "Mavyret treatment" arm will not be comparable groups with regard to the outcomes of this study.

#### 10.4.7 Planned Interim Analysis

Interim analysis not applicable

#### 10.4.7.1 Safety Review

Any patient death will result in halting of any further enrollment in the study and an assessment of whether the death was related to HCV exposure, infection, or treatment. Even in the event of a patient death, currently enrolled patients who are actively being treated for HCV viremia and tolerating therapy will continue to receive therapy so as not to put them at risk for HCV infection and/or the development of resistance as a consequence of interrupted therapy. If the patient death is deemed related to a specific treatment agent, enrolled patients receiving that same agent will be switched to an alternative therapy.

#### 10.4.8 Multiple Comparison/Multiplicity

Not applicable.

#### 10.4.9 Tabulation of Individual Response Data

Since this is a relatively small trial, individual participant data, in particular as pertains to the kinetics of the development and clearance of HCV viremia, will be evaluated.


# 10.5 Sample Size

10 patients are expected to enroll in this trial.

We expect that less approximately 70% of patients will develop evidence of HCV infection transmitted from the HCV-positive donor and will be treated for HCV infection. We expect that 100% of the patients who are treated for HCV infection will achieve SVR.

This is a single-arm study with no comparison group. The power to detect a difference in observed versus expected depends upon the true efficacy of the therapy. The reported efficacy of the therapy is 98%. With an estimated 7 patients who will be treated, a single treatment failure will be regarded as a significant deviation from the expected outcome.

#### 11 Source Documents and Access to Source Data/Documents

Source data is all information, original records of clinical findings, observations, or other activities in a clinical trial necessary for the reconstruction and evaluation of the trial. Source data are contained in source documents. Examples of these original documents, and data records include: hospital records, clinical and office charts, laboratory notes, memoranda, subjects' diaries or evaluation checklists, pharmacy dispensing records, recorded data from automated instruments, copies or transcriptions certified after verification as being accurate and complete, microfiches, photographic negatives, microfilm or magnetic media, x-rays, subject files, and records kept at the pharmacy, at the laboratories, and at medico-technical departments involved in the clinical trial. It is acceptable to use CRFs as source documents. If this is the case, it should be stated in this section what data will be collected on CRFs and what data will be collected from other sources.

The study case report form (CRF) is the primary data collection instrument for the study. All data requested on the CRF must be recorded. All missing data must be explained. If a space on the CRF is left blank because the procedure was not done or the question was not asked, write "N/D". If the item is not applicable to the individual case, write "N/A". All entries should be printed legibly in black ink. If any entry error has been made, to correct such an error, draw a single straight line through the incorrect entry and enter the correct data above it. All such changes must be initialed and dated. DO NOT ERASE OR WHITE OUT ERRORS. For clarification of illegible or uncertain entries, print the clarification above the item, then initial and date it.

Access to study records will be limited to IRB-approved members of the study team. The investigator will permit study-related monitoring, audits, and inspections by the IRB/EC, the sponsor, government regulatory bodies, and University compliance and quality assurance groups of all study related documents (e.g. source documents, regulatory documents, data collection instruments, study data etc.). The investigator will ensure the capability for inspections of applicable study-related facilities (e.g. pharmacy, diagnostic laboratory, etc.).

Participation as an investigator in this study implies acceptance of potential inspection by government regulatory authorities and applicable University compliance and quality assurance offices.

#### 12 Quality Assurance and Quality Control

QC procedures will be implemented beginning with the data entry system and data QC checks that will be run on the database will be generated. Any missing data or data anomalies will be communicated to the site(s) for clarification/resolution.

Following written SOPs, the monitors will verify that the clinical trial is conducted and data are generated, documented (recorded), and reported in compliance with the protocol, GCP, and the applicable regulatory requirements (e.g., Good Laboratory Practices (GLP), Good Manufacturing Practices (GMP)).


The investigational site will provide direct access to all trial related sites, source data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and regulatory authorities.

#### 13 Ethics/Protection of Human Subjects

#### 13.1 Ethical Standard

The investigator will ensure that this study is conducted in full conformity with Regulations for the Protection of Human Subjects of Research codified in 45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, and/or the ICH E6.

#### 13.2 Institutional Review Board

The protocol, informed consent form, recruitment materials, and all participant materials will be submitted to the IRB for review and approval. Approval of both the protocol and the consent form must be obtained before any participant is enrolled. Any amendment to the protocol will require review and approval by the IRB before the changes are implemented to the study. All changes to the consent form will be IRB approved; a determination will be made regarding whether previously consented participants need to be re-consented.

#### 13.3 Informed Consent Process

#### 13.3.1 Consent/Assent and Other Informational Documents Provided to Participants

Consent forms describing in detail the study agent, study procedures, and risks are given to the participant and written documentation of informed consent is required prior to starting intervention/administering study product. The informed consent document to be used is submitted with this protocol.

#### 13.3.2 Consent Procedures and Documentation

Informed consent is a process that is initiated prior to the individual's agreeing to participate in the study and continues throughout the individual's study participation. Extensive discussion of risks and possible benefits of participation will be provided to the participants and their families. Consent forms will be IRB-approved and the participant will be asked to read and review the document. The investigator will explain the research study to the participant and answer any questions that may arise. All participants will receive a verbal explanation in terms suited to their comprehension of the purposes, procedures, and potential risks of the study and of their rights as research participants. Participants will have the opportunity to carefully review the written consent form and ask questions prior to signing. The participants should have the opportunity to discuss the study with their surrogates or think about it prior to agreeing to participate. The participant will sign the informed consent document prior to any procedures being done specifically for the study. The participants may withdraw consent at any time throughout the course of the trial. A copy of the signed informed consent document will be given to the participants for their records. The rights and welfare of the participants will be protected by emphasizing to them that the quality of their medical care will not be adversely affected if they decline to participate in this study.

A copy of the signed informed consent document will be stored in the subject's research record. The consent process, including the name of the individual obtaining consent, will be thoroughly documented in the subject's research record. Any alteration to the standard consent process (e.g. use of a translator,


consent from a legally authorized representative, consent document presented orally, etc.) and the justification for such alteration will likewise be documented.

#### 13.4 Participant and Data Confidentiality

Information about study subjects will be kept confidential and managed according to the requirements of the Health Insurance Portability and Accountability Act of 1996 (HIPAA). Those regulations require a signed subject authorization informing the subject of the following:

- What protected health information (PHI) will be collected from subjects in this study
- Who will have access to that information and why
- Who will use or disclose that information
- The rights of a research subject to revoke their authorization for use of their PHI.

In the event that a subject revokes authorization to collect or use PHI, the investigator, by regulation, retains the ability to use all information collected prior to the revocation of subject authorization. For subjects that have revoked authorization to collect or use PHI, attempts should be made to obtain permission to collect at least vital status (i.e. that the subject is alive) at the end of their scheduled study period.

Participant confidentiality is strictly held in trust by the participating investigators, their staff, and the sponsor(s) and their agents. This confidentiality is extended to cover testing of biological samples and genetic tests in addition to the clinical information relating to participants. Therefore, the study protocol, documentation, data, and all other information generated will be held in strict confidence. No information concerning the study or the data will be released to any unauthorized third party without prior written approval of the sponsor.

The study monitor, other authorized representatives of the IRB may inspect all documents and records required to be maintained by the investigator, including but not limited to, medical records (office, clinic, or hospital) and pharmacy records for the participants in this study. The clinical study site will permit access to such records.

The study participant's contact information will be securely stored at each clinical site for internal use during the study. At the end of the study, all records will continue to be kept in a secure location for as long a period as dictated by local IRB and Institutional regulations.

Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored at NYU Langone Medical Center. This will not include the participant's contact or identifying information. Rather, individual participants and their research data will be identified by a unique study identification number. The study data entry and study management systems used by clinical sites and by NYU Langone Medical Center research staff will be secured and password protected. At the end of the study, all study databases will be de-identified and archived at the NYU Langone Medical Center.

#### 14 Data Handling and Record Keeping

#### 14.1 Data Collection and Management Responsibilities

Data collection is the responsibility of the clinical trial staff at the site under the supervision of the site PI. The investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported.

All source documents should be completed in a neat, legible manner to ensure accurate interpretation of data. Black ink is required to ensure clarity of reproduced copies. When making changes or corrections,


This material is the property of the NYU School of Medicine and Langone Medical Center. Do not disclose or use except as authorized in writing by the study sponsor


cross out the original entry with a single line, and initial and date the change. DO NOT ERASE, OVERWRITE, OR USE CORRECTION FLUID OR TAPE ON THE ORIGINAL.

Data will be collected on CRFs and maintained in the study binder. Copies of the CRF will be provided for use as source documents and maintained for recording data for each participant enrolled in the study. Data reported in the CRF derived from source documents should be consistent with the source documents or the discrepancies should be explained and captured in a progress note and maintained in the participant's official electronic study record.

Clinical data (including AEs, concomitant medications, and expected adverse reactions data) and clinical laboratory data will be assimilated in the study subject binders. Clinical data will be entered directly from the source documents.

# 14.2 Study Records Retention

Study documents will be retained for the longer of 3 years after close-out, 5 years after final reporting/publication, or 2 years after the investigation is discontinued. No records will be destroyed without the written consent of the sponsor, if applicable. It is the responsibility of the sponsor to inform the investigator when these documents no longer need to be retained.

#### 14.3 Protocol Deviations

A protocol deviation is any noncompliance with the clinical trial protocol, GCP, or Manual of Procedures (MOP) requirements. The noncompliance may be either on the part of the participant, the investigator, or the study site staff. As a result of deviations, corrective actions are to be developed by the site and implemented promptly.

These practices are consistent with ICH E6:

- 4.5 Compliance with Protocol, sections 4.5.1, 4.5.2, and 4.5.3
- 5.1 Quality Assurance and Quality Control, section 5.1.1
- 5.20 Noncompliance, sections 5.20.1, and 5.20.2.

It is the responsibility of the site PI/study staff to use continuous vigilance to identify and report deviations within 3 working days of identification of the protocol deviation, or within 3 working days of the scheduled protocol-required activity.

All protocol deviations must be addressed in study source documents, reported to the Monitoring committee and the IRB.

Protocol deviations must be reported to the local IRB per their guidelines. The site PI/study staff is responsible for knowing and adhering to their IRB requirements. Further details about the handling of protocol deviations will be included in the MOP.

## 14.4 Publication and Data Sharing Policy

This study will comply with the NIH Public Access Policy, which ensures that the public has access to the published results of NIH funded research. It requires scientists to submit final peer-reviewed journal manuscripts that arise from NIH funds to the digital archive PubMed Central upon acceptance for publication.

The International Committee of Medical Journal Editors (ICMJE) member journals have adopted a clinical trials registration policy as a condition for publication. The ICMJE defines a clinical trial as any research CONFIDENTIAL

This material is the property of the NYU School of Medicine and Langone Medical Center. Do not disclose or use except as authorized in writing by the study sponsor


project that prospectively assigns human subjects to intervention or concurrent comparison or control groups to study the cause-and-effect relationship between a medical intervention and a health outcome. Medical interventions include drugs, surgical procedures, devices, behavioral treatments, process-of-care changes, and the like. Health outcomes include any biomedical or health-related measures obtained in patients or participants, including pharmacokinetic measures and adverse events. The ICMJE policy, and the Section 801 of the Food and Drug Administration Amendments Act of 2007, requires that all clinical trials be registered in a public trials registry such as ClinicalTrials.gov, which is sponsored by the National Library of Medicine. Other biomedical journals are considering adopting similar policies. For interventional clinical trials performed under NIH IC grants and cooperative agreements, it is the grantee's responsibility to register the trial in an acceptable registry, so the research results may be considered for publication in ICMJE member journals. The ICMJE does not review specific studies to determine whether registration is necessary; instead, the committee recommends that researchers who have questions about the need to register err on the side of registration or consult the editorial office of the journal in which they wish to publish.

FDAAA mandates that a "responsible party" (i.e., the sponsor or designated principal investigator) register and report results of certain "applicable clinical trials":

- Trials of Drugs and Biologics: Controlled, clinical investigations, other than Phase I investigations of a product subject to FDA regulation;
- Trials of Devices: Controlled trials with health outcomes of a product subject to FDA regulation (other than small feasibility studies) and pediatric postmarket surveillance studies.
- NIH grantees must take specific steps to ensure compliance with NIH implementation of FDAAA.

## 15 Study Finances

## 15.1 Funding Source

Medication costs for the study drug Mavyret will be paid by the Transplant Institute. Study specific laboratory testing will be limited to:

- Serial HCV PCR and serology testing which will be performed at a greater frequency than for standard of care following heart transplantation.
- Genotyping of donor HCV
- Genotyping of recipient HCV among those who develop viremia

The costs of these laboratory tests will be covered by the Transplant Institute.

All other medications and laboratory testing required for this study are routinely conducted as standard of care for all recipients of heart transplants and are not considered components of the study.

## 15.2 Costs to the Participant

Participants will not incur any costs associated with participating in this trial.

## 16 Study Administration

### 16.1 Study Leadership

The Principal Investigator will govern the conduct of the study. The PI, together with at least one coinvestigator will meet in person or by teleconference with the DSMB (at least 4 members) at least quarterly and documentation of the meeting will be maintained.

## 17 Conflict of Interest Policy

The independence of this study from any actual or perceived influence, such as by the pharmaceutical industry, is critical. Therefore, any actual conflict of interest of persons who have a role in the design,

## CONFIDENTIAL

This material is the property of the NYU School of Medicine and Langone Medical Center. Do not disclose or use except as authorized in writing by the study sponsor


conduct, analysis, publication, or any aspect of this trial will be disclosed and managed. Furthermore, persons who have a perceived conflict of interest will be required to have such conflicts managed in a way that is appropriate to their participation in the trial. The study leadership in conjunction with NYULMC has established policies and procedures for all study group members to disclose all conflicts of interest and will establish a mechanism for the management of all reported dualities of interest.

Any investigator who has a conflict of interest with this study (patent ownership, royalties, or financial gain greater than the minimum allowable by their institution, etc.) must have the conflict reviewed by the NYU Langone Conflict of Interest Management Unit (CIMU) with a Committee-sanctioned conflict management plan that has been reviewed and approved by the study sponsor prior to participation in this study. All NYULMC investigators will follow the applicable conflict of interest policies.


#### 18 References

- 1. Organ Procurement and Transplantation Network (OPTN) https://optn.transplant.hrsa.gov
- 2. Lonze B.E., Unpublished analyses of data provided by the Scientific Registry of Transplant Recipients (SRTR).
- 3. Alkhouri, N., E. Lawitz, and F. Poordad, *Novel treatments for chronic hepatitis C: closing the remaining gaps*. Curr Opin Pharmacol, 2017. **37**: p. 107-111.
- 4. Goldberg, D.S., et al., *Trial of Transplantation of HCV-Infected Kidneys into Uninfected Recipients*. N Engl J Med, 2017. **376**(24): p. 2394-2395.
- 5. Desai, N. N., The Johns Hopkins Hospital, personal communication.
- 6. Shah, A.S., Vanderbilt University Hospital, personal communication.
- 7. Levitsky, J., et al., *The American Society of Transplantation Consensus Conference on the Use of Hepatitis C Viremic Donors in Solid Organ Transplantation*. Am J Transplant, 2017. **17**(11): p. 2790-2802.
- 8. Ng, T.I., et al., *In Vitro Antiviral Activity and Resistance Profile of the Next-Generation Hepatitis C Virus NS3/4A Protease Inhibitor Glecaprevir.* Antimicrob Agents Chemother, 2017.
- 9. Asselah, T., et al., Efficacy of Glecaprevir/Pibrentasvir for 8 or 12 Weeks in Patients With Hepatitis C Virus Genotype 2, 4, 5, or 6 Infection Without Cirrhosis. Clin Gastroenterol Hepatol, 2017.
- 10. Forns, X., et al., Glecaprevir plus pibrentasvir for chronic hepatitis C virus genotype 1, 2, 4, 5, or 6 infection in adults with compensated cirrhosis (EXPEDITION-1): a single-arm, open-label, multicentre phase 3 trial. Lancet Infect Dis, 2017. **17**(10): p. 1062-1068.
- 11. Hubbard, H. and E. Lawitz, *Glecaprevir + pibrentasvir (ABT493 + ABT-530) for the treatment of Hepatitis C.* Expert Rev Gastroenterol Hepatol, 2017: p. 1-9.
- 12. Kumada, H., et al., Efficacy and safety of glecaprevir/pibrentasvir in HCV-infected Japanese patients with prior DAA experience, severe renal impairment, or genotype 3 infection. J Gastroenterol, 2017.
- 13. Kwo, P.Y., et al., Glecaprevir and pibrentasvir yield high response rates in patients with HCV genotype 1-6 without cirrhosis. J Hepatol, 2017. **67**(2): p. 263-271.
- 14. Poordad, F., et al., *Glecaprevir/Pibrentasvir in Patients with HCV Genotype 1 or 4 and Prior Direct-acting Antiviral Treatment Failure*. Hepatology, 2017.
- 15. Gane, E., et al., *Glecaprevir and Pibrentasvir in Patients with HCV and Severe Renal Impairment.* N Engl J Med, 2017. **377**(15): p. 1448-1455.
- 16. HCV Guidance: Recommendations for Testing, Managing, and Treating Hepatitis C.
- 17. AbbVie, Inc., Mavyret, presribing information.
- 18. Farci, P., et al., *Hepatitis C virus-associated fulminant hepatic failure.* N Engl J Med, 1996. **335**(9): p. 631-4.
- 19. Dustin, L.B., *Innate and Adaptive Immune Responses in Chronic HCV Infection.* Curr Drug Targets, 2017. **18**(7): p. 826-843.
- 20. Singh, T.P., et al., Survival benefit from transplantation in patients listed for heart transplantation in the United States. J Am Coll Cardiol, 2014. **63**(12): p. 1169-1178.


# 19 Attachments

These documents are relevant to the protocol, but they are not considered part of the protocol. On the following two pages are:

- Sample Study Fact Sheet
- Sample of Acknowledgment of Willingness to Participate Form

The following additional documents relevant to this study can be founds as uploads in the Research Navigator:

- SOP for specimen handling
- Accreditation letter for the Transplant Laboratory
- Specimen collection and shipping instructions for Quest Diagnostics


Study#: s17-01775 Version date: 17 December 2017

Page 1 of 1



# **HCV Heart Research Study Fact Sheet**

**Title of Study:** A single-center pilot study of the use of hepatitis C positive donors for hepatitis

C negative hear transplant with post-transplant treatment of hepatitis C

viremia with Mavyret

IRB study number: s17-01775

Principal Investigator:

Alex Reyentovich, MD Department of Medicine NYU School of Medicine

530 First Avenue, Skirball 9V, New York, NY 10016

Because you are being evaluated as a candidate for a heart transplant, you may qualify to participate in the abovenamed research study. Participation in the study is voluntary. Your interest in this study will not affect your placement on the waiting list, or your position on the waiting list.

This study is being done because there is a shortage of organ donors for heart transplants, and many patients die while on the waiting list for a heart transplant.

Hearts from donors who test positive for hepatitis C (HCV) are currently discarded and not used for transplant. Using these hearts would potentially eliminate the organ shortage problem. This would reduce the waiting list, and would reduce the risk of death on the waiting list.

In this study, hearts from donors who test positive for HCV infection will be transplanted into patients who are negative for HCV. By receiving a transplant from a HCV donor, there is a possibility that you will be exposed to HCV or infected with HCV.

There are readily available treatments for HCV that can cure HCV infection with a success rate of over 95%. Patients in this study will have frequent blood tests after transplant to determine whether any HCV infection has occurred. Patients who develop HCV infection after transplant will receive treatment with an FDA-approved drug that is effective in the treatment of all types of HCV. The drug is called MAVYRET.

Participation in the study would last about 12 months from the time of the transplant. Participation will involve weekly blood tests to check for HCV infection after transplant. If HCV infection is found, the treatment will be a medication called MAVYRET that is taken by mouth every day for 8 weeks. This medication will be provided at no cost to you. Once the treatment is completed, there will be additional regular lab tests to ensure that the infection has cleared. Patients who do not develop HCV infection will not be treated with MAVYRET.

The most important risk of this study would be if HCV infection is not able to be cured with treatment, you could develop liver disease and, rarely, liver failure requiring a liver transplant. We think these risks are low.

The most important benefits of this study are that accepting a heart from a HCV positive donor will enable you to get a heart transplant more quickly, and that this will reduce your chances of dying on the waiting list.


Study #: s17-01775 Version date: 17 December 2017

Page 1 of 1



# Potential Research Subject Willingness to Participate Form

Title of Study: A single-center pilot study of the use of hepatitis C positive donors for hepatitis

C negative hear transplant with post-transplant treatment of hepatitis C

viremia with Mavyret.

IRB study number: s17-01775

Principal Investigator:

Alex Reyentovich, MD Department of Medicine NYU School of Medicine

530 First Avenue, Skirball 9V, New York, NY 10016

## This form does NOT constitute consent to enroll in the above study.

By signing this form, I acknowledge that I have been informed that participation in the above study may be an option for me. The potential risks and benefits of this study have been explained to me and I have received a copy of the HCV Heart Research Study Fact Sheet.

Signing this form does not guarantee that I will be enrolled in this study.

Signing this form does not mean that I cannot receive a heart transplant at NYU Langone outside of this study.

Signing this form designates that if a suitable organ offer from an HCV positive heart donor becomes available, I would like to be contacted and offered enrollment in the study.

| Name of Patient (Print) | Signature of Patient | Date |
|---|---|---|
| Marno of Domon Droviding this Form (Drint) | Cinnatura of Doman Draviding this Form | Dato |

# 20 Schedule of Events

For patients who do not develop HCV viremia during the surveillance phase, the following schedule will apply for the entire course of the study:

| Activity | Screening visit<br>(Day -365 to -1) | Enrollment | SURVEILLANCE PHASE | | | |
|---|---|---|---|---|---|---|
| | | visit | POW1 | POW2 | POW3 | POW4 |
| | | (Day -1 to 0) | (+/- 1 day) | (+/- 2 day) | (+/- 3 day) | (+/- 5 day) |
| Study team procedures | | | | | | |
| Acknowledgement of willingness to participate, provision of Study Fact Sheet | X | | | | | |
| Medical History | X | | | | | |
| Physical Exam | X | Χ | X | Χ | | |
| Height | X | X | X | X | | X |
| Weight | X | Х | Х | X | | Х |
| Vitals signs | Х | Х | Х | Х | | Х |
| Review all donor and recipient inclusion/exclusion criteria | | Х | | | | |
| Signing of informed consent | | X | | | | |
| Study specific interventions | | | | | | |
| Heart transplant operation | | Х | | | | |
| Initiate Mavyret treatment | | | | | | |
| Study specific laboratory tests | | | | | | |
| Donor serum HCV genotyping | | Х | | | | |
| Recipient serum HCV genotyping | | | | | | |
| HCV NAT (PCR) | Х | Х | Х | Х | Х | Х |
| HCV serology (HCV Ab) | Х | Х | | | | |
| SOC laboratory tests | | | | | | |
| Biochemistry (Na, K, CO2, BUN, Cr, total bili, AST, ALT, alk phos) | Х | Х | Х | Х | Х | Х |
| Hematology (WBC with ANC, HGB, PLT) | X | X | Х | X | X | Х |
| Coagulation (INR) | Х | Х | Х | Х | Х | Х |
| Urine pregnancy test | | Х | | | | |
| HBV NAT (PCR) | Х | Х | | | | |
| HBV serology (HBsAb, HBsAg, HBcoreAb) | Х | Х | | | | |
| HIV serology (HIV1/2 antigen/antibody 4 <sup>th</sup> gen) | Х | Х | | | | |

| Activity | | SURVEILLA | POW12 | POW16 | | |
|---|---|---|---|---|---|---|
| | <b>POW5</b> (+/- 5 days) | <b>POW6</b> (+/- 5 days) | <b>POW7</b> (+/- 5 days) | <b>POW8</b> (+/- 5 days) | (+/- 7 days) | (+/- 7 days) |
| Study team procedures | | | | | | |
| Acknowledgement of willingness to participate, provision of Study Fact Sheet | | | | | | |
| Medical History | | | | | | |
| Physical Exam | | | | | | |
| Height | | | | Х | Х | |
| Weight | | | | Х | Х | |
| Vitals signs | | | | Х | Х | |
| Review all donor and recipient inclusion/exclusion criteria | | | | | | |
| Signing of informed consent | | | | | | |
| Study specific interventions | | | | | | |
| Heart transplant operation | | | | | | |
| Initiate Mavyret treatment | | | | | | |
| Study specific laboratory tests | | | | | | |
| Donor serum HCV genotyping | | | | | | |
| Recipient serum HCV genotyping | | | | | | |
| HCV NAT (PCR) | Х | Х | X | Х | Х | Х |
| HCV serology (HCV Ab) | | | | Х | Х | Х |
| SOC laboratory tests | | | | | | |
| Biochemistry (Na, K, CO2, BUN, Cr, total bili, AST, ALT, alk phos) | Х | Х | Х | Х | Х | Х |
| Hematology (WBC with ANC, HGB, PLT) | Х | Х | Х | Х | Х | Х |
| Coagulation (INR) | Х | Х | Х | Х | Х | Х |
| Urine pregnancy test | | | | | | |
| HBV NAT (PCR) | | | | | Х | |
| HBV serology (HBsAb, HBsAg, HBcoreAb) | | | | | Х | |
| HIV serology (HIV1/2 antigen/antibody 4 <sup>th</sup> gen) | | | | | Х | |

| Activity | <b>POW20</b> (+/- 7 days) | POW 24 - Interim<br>assessment visit<br>(+/- 14 days) | POW 52 - Final<br>assessment visit<br>(+/- 14 days) |
|---|---|---|---|
| Study team procedures | | · · · · · | |
| Acknowledgement of willingness to participate, provision of Study Fact Sheet | | | |
| Medical History | | | |
| Physical Exam | | | |
| Height | | | X |
| Weight | | | X |
| Vitals signs | | | X |
| Review all donor and recipient inclusion/exclusion criteria | | | |
| Signing of informed consent | | | |
| Study specific interventions | | | |
| Heart transplant operation | | | |
| Initiate Mavyret treatment | | | |
| Study specific laboratory tests | | | |
| Donor serum HCV genotyping | | | |
| Recipient serum HCV genotyping | | | |
| HCV NAT (PCR) | Х | Χ | X |
| HCV serology (HCV Ab) | Х | Х | Х |
| SOC laboratory tests | | | |
| Biochemistry (Na, K, CO2, BUN, Cr, total bili, AST, ALT, alk phos) | Х | Х | Х |
| Hematology (WBC with ANC, HGB, PLT) | X | Χ | X |
| Coagulation (INR) | X | Χ | X |
| Urine pregnancy test | | | |
| HBV NAT (PCR) | | | Х |
| HBV serology (HBsAb, HBsAg, HBcoreAb) | | | X |
| HIV serology (HIV1/2 antigen/antibody 4 <sup>th</sup> gen) | | | X |

| Activity | MAVYRET TREATMENT PHASE | | | | | |
|---|---|---|---|---|---|---|
| | <b>PMW0</b> (+/- 5 days) | <b>PMW1</b> (+/- 1 day) | <b>PMW2</b> (+/- 2 days) | <b>PMW3</b> (+/- 3 days) | <b>PMW4</b> (+/- 5 days) | <b>PMW5</b> (+/- 5 days) |
| Study team procedures | | | | | | |
| Acknowledgement of willingness to participate, provision of Study Fact Sheet | | | | | | |
| Medical History | | | | | | |
| Physical Exam | Х | | | | | |
| Height | Х | | | | Х | |
| Weight | Х | | | | Х | |
| Vitals signs | Х | | | | Х | |
| Review all donor and recipient inclusion/exclusion criteria | | | | | | |
| Signing of informed consent | | | | | | |
| Study specific interventions | | | | | | |
| Heart transplant operation | | | | | | |
| Initiate Mavyret treatment | Х | | | | | |
| Study specific laboratory tests | | | | | | |
| Donor serum HCV genotyping | | | | | | |
| Recipient serum HCV genotyping | Х | | | | | |
| HCV NAT (PCR) | | Х | Х | X | Х | Х |
| HCV serology (HCV Ab) | | Х | Х | Х | Х | Х |
| SOC laboratory tests | | | | | | |
| Biochemistry (Na, K, CO2, BUN, Cr, total bili, AST, ALT, alk phos) | | Х | Х | Х | Х | Х |
| Hematology (WBC with ANC, HGB, PLT) | | Х | Х | X | Х | Х |
| Coagulation (INR) | | Х | Х | Х | Х | Х |
| Urine pregnancy test | | | | | | |
| HBV NAT (PCR) | | | | | | |
| HBV serology (HBsAb, HBsAg, HBcoreAb) | | | | | | |
| HIV serology (HIV1/2 antigen/antibody 4 <sup>th</sup> gen) | | | | | | |

| | MAVYRET TREATMENT PHASE | | | PMW9 | PMW10 | PMW11 |
|---|---|---|---|---|---|---|
| Activity | PMW6 | PMW7 | PMW8 | (+/- 5 days) | (+/- 5 days) | (+/- 5 days) |
| | (+/- 5 days) | (+/- 5 days) | (+/- 5 days) | , , | , , | |
| Study team procedures | | | | | | |
| Acknowledgement of willingness to participate, provision of Study Fact Sheet | | | | | | |
| Medical History | | | | | | |
| Physical Exam | | | | | | |
| Height | | | Х | | | |
| Weight | | | Х | | | |
| Vitals signs | | | Х | | | |
| Review all donor and recipient inclusion/exclusion criteria | | | | | | |
| Signing of informed consent | | | | | | |
| Study specific interventions | | | | | | |
| Heart transplant operation | | | | | | |
| Initiate Mavyret treatment | | | | | | |
| Study specific laboratory tests | | | | | | |
| Donor serum HCV genotyping | | | | | | |
| Recipient serum HCV genotyping | | | | | | |
| HCV NAT (PCR) | X | X | X | X | X | Х |
| HCV serology (HCV Ab) | X | X | X | X | X | Х |
| SOC laboratory tests | | | | | | |
| Biochemistry (Na, K, CO2, BUN, Cr, total bili, AST, ALT, alk phos) | Х | Х | Х | Х | Х | Х |
| Hematology (WBC with ANC, HGB, PLT) | X | X | X | X | X | X |
| Coagulation (INR) | Х | X | Х | X | Х | Х |
| Urine pregnancy test | | | | | | |
| HBV NAT (PCR) | | | | | | |
| HBV serology (HBsAb, HBsAg, HBcoreAb) | | | | | | |
| HIV serology (HIV1/2 antigen/antibody 4 <sup>th</sup> gen) | | | | | | |

| Activity | <b>PMW12</b> (+/- 5 days) | <b>PMW16</b> (+/- 7 days) | POW 24 - Interim<br>assessment visit<br>(+/- 14 days) | POW 52 - Final<br>assessment visit<br>(+/- 14 days) |
|---|---|---|---|---|
| Study team procedures | | | | |
| Acknowledgement of willingness to participate, provision of Study Fact Sheet | | | | |
| Medical History | | | | |
| Physical Exam | | | | |
| Height | | | | X |
| Weight | | | | X |
| Vitals signs | | | | Х |
| Review all donor and recipient inclusion/exclusion criteria | | | | |
| Signing of informed consent | | | | |
| Study specific interventions | | | | |
| Heart transplant operation | | | | |
| Initiate Mavyret treatment | | | | |
| Study specific laboratory tests | | | | |
| Donor serum HCV genotyping | | | | |
| Recipient serum HCV genotyping | | | | |
| HCV NAT (PCR) | Х | X | X | Х |
| HCV serology (HCV Ab) | Х | X | Х | Х |
| SOC laboratory tests | | | | |
| Biochemistry (Na, K, CO2, BUN, Cr, total bili, AST, ALT, alk phos) | Х | × | Х | Х |
| Hematology (WBC with ANC, HGB, PLT) | Х | X | Х | X |
| Coagulation (INR) | Х | Х | Х | X |
| Urine pregnancy test | | | | |
| HBV NAT (PCR) | | | | X |
| HBV serology (HBsAb, HBsAg, HBcoreAb) | | | | X |
| HIV serology (HIV1/2 antigen/antibody 4 <sup>th</sup> gen) | | | | X |